CLINICAL TRIAL: NCT05948449
Title: The Efficacy and Safety of Chemotherapy Combined With Cadonilimab (AK104) in Neoadjuvant Treatment of Locally Advanced Gastric Cancer/Gastroesophageal Junction Adenocarcinoma: A Prospective, Single-arm, Phase II Clinical Study
Brief Title: To Evaluate the Efficacy and Safety of Cadonilimab With SOX as Neoadjuvant Therapy for Resectable Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Director, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH-2023-526
Record Dates: First submitted 2023-07-10; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; neoadjuvant therapy; Cadonilimab
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOX+Cadonilimab（AK104） (Experimental): 3 cycles of neoadjuvant therapy: S-1: 40~60mg Bid，d1~14, q3w Oxaliplatin：130mg/m2，iv drip，d1, q3w Cadonilimab（AK104）:10mg/Kg,iv drip,d1,q3w
  Interventions: Drug: S-1, Oxaliplatin, Cadonilimab

INTERVENTIONS:
Drug: S-1, Oxaliplatin, Cadonilimab — 3 cycles of neoadjuvant therapy will be administered: S-1: 40~60mg Bid，d1~14, q3w Oxaliplatin：130mg/m2，iv drip，d1, q3w Cadonilimab（AK104）:10mg/Kg,iv drip,d1,q3w

SUMMARY:
The Purpose of This Study is to Evaluate the Efficacy and Safety of Cadonilimab（AK104） in Combination With SOX as Neoadjuvant Therapy for Patients With Resectable Locally Advanced Gastric or Gastroesophageal Adenocarcinoma.

DETAILED DESCRIPTION:
Recent years, neoadjuvant therapy have emerged as a promising treatment option for the treatment of locally advanced gastric or gastroesophageal adenocarcinoma. However, the efficacy of current neoadjuvant regimens is still unsatisfactory. Novel treatment with higher efficacy and safety are urgently needed. Recently, immunotherapy has achieved significant therapeutic effects in the treatment of a series of cancers, and chemotherapy combined with immunotherapy has been recommended as the standard first-line treatment for gastric cancer. Moreover, several phase I/II studies have explored the efficacy and safety of chemotherapy combined with PD-1 inhibitor in the neoadjuvant treatment for gastric cancer, the results of which indicate that chemotherapy combined with immunotherapy can significantly improve the pCR rate and R0 resection rate of gastric cancer. In this study, we will evaluate the efficacy and safety of chemotherapy combined with Cadonilimab（AK104） (a PD-1/CTLA-4 bispecific antibody) in the neoadjuvant therapy for resectable locally advanced gastric or gastroesophageal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Histologically or cytologically confirmed diagnosis of adenocarcinoma locate at gastroesophageal junction or stomach, advanced gastric or gastroesophageal junction cancer as assessed by ultrasonography and/or CT/MRI (cT3-T4a, N+, M0).
3. Resectable gastric or gastroesophageal cancer, judged by surgeons in this study.
4. No previous anti-tumor treatment.
5. The expected survival is no less than 3 months.
6. ECOG PS≤1.
7. Adequate organ function including the following:

   * Total bilirubin ≤1.5 times upper limit of normal (ULN),
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3×ULN,
   * Alkaline phosphatase≤2.5×ULN (If the tumor invaded the liver, ≤3×ULN),
   * Serum creatinine≤1.5×ULN,
   * Serum amylase and lipase≤1.5×ULN,
   * International standardized ratio (INR)/partial prothrombin time (PTT)≤1.5×ULN;
   * Platelet count ≥ 75,000 /mm3.
   * Hemoglobin (Hb) ≥ 9 g/dL.
   * Absolute neutrophil count (ANC) ≥ 1500/mm3.
8. Strict contraception.
9. Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

1. Unable to comply with the research program or procedures.
2. Undergoing other drug clinical trials, or has participated in any drug clinical trials one month before enrollment.
3. Active autoimmune disease or history of refractory autoimmune disease.
4. Receiving corticosteroid (> 10mg/d prednisone or equivalent dose of steroids) or other systematic immunosuppression therapies within 14 days before enrollment, excluding following therapies: steroid hormone replacement therapy (≤10mg/d); local steroid therapy; short-term, prophylactic steroid therapy for preventing allergies or nausea and vomiting.
5. Active or clinically significant cardiac disease:

   * Congestive heart failure > New York Heart Association (NYHA ) class 2;
   * Active coronary artery disease;
   * Arrhythmias requiring treatment other than β-blocker or digoxin;
   * Unstable angina (with angina symptoms at rest), new angina within 3 months before enrollment, or new myocardial infarction within 6 months before enrollment
6. Evidence or history of bleeding diathesis or coagulopathy.
7. Grade 3 bleeding events 4 weeks before enrollment.
8. Thromboembolism or arteriovenous events, such as cerebrovascular events (including transient ischemic attack), deep vein thrombosis or pulmonary embolism, occurred 6 months before enrollment.
9. Currently taking anticoagulants.
10. Other tumors that have not been treated or exist at the same time, except carcinoma in situ of the cervix, treated basal cell carcinoma or superficial bladder tumor. If the tumor has been cured and no evidence of disease has been found for more than 3 years, the patient can be enrolled. All other tumors must be treated at least 3 years before enrollment.
11. Patients with pheochromocytoma.
12. Patients with a history of HIV infection or active hepatitis B/C.
13. Ongoing > level 2 infection.
14. Symptomatic brain metastasis or meningioma.
15. Unhealed wounds, ulcers or fractures.
16. Renal failure patients requiring blood or peritoneal dialysis.
17. Dehydration≥ 1 grade.
18. Epileptic that need medication.
19. Active, symptomatic interstitial pneumonia, pleural or ascites that causes dyspnea (dyspnea ≥ 2 grade).
20. History of organ transplantation. (including corneal transplantation).
21. Allergic to research drugs or similar drugs, or suspected allergies.
22. Malabsorption patients.
23. Pregnant or lactating women.
24. Investigator believes that patients who are not suitable for the study.
25. Medical, psychological or social conditions can affect the recruitment of patients and evaluation for study results.
26. Other anti-tumor therapy (chemotherapy, radiotherapy, surgery, immunotherapy, biotherapy, chemoembolization) other than investigator drugs. Palliative external irradiation for non-target lesions is allowed.
27. Previously used oxaliplatin, S-1 or Cadonilimab.
28. Major surgery 4 weeks before recruitment, open biopsy or major trauma surgery. (excluding biliary stents, or percutaneous biliary drainage).
29. Treatment with anti-tumor Chinese herbal medicine.
30. History of allogeneic blood transfusion within 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  evaluate pathological complete response rate of primary tumor and locally metastatic lymph nodes after 3 cycles of neoadjuvant therapy.

SECONDARY OUTCOMES:
R0 resection rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Rate of microscopically margin-negative resection
2-year overall survival rate | 2 years
2-year disease free survival rate | 2 year
major pathological response (MPR) | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
Safety and Tolerability | 3 months after the last administration of drugs
  Treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jiankun Hu, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang PF, Zhang WH, Liu XJ, He D, Yang K, Gou HF, Hu JK. Chemotherapy combined with cadonilimab (AK104) as neoadjuvant treatment for locally advanced gastric/gastro-oesophageal junction adenocarcinoma: study protocol for a single-arm, phase II clinical trial. BMJ Open. 2024 Dec 4;14(12):e081529. doi: 10.1136/bmjopen-2023-081529. PMID 39632107